CLINICAL TRIAL: NCT00623935
Title: Hematopoietic Stem Cell Transplantation for the Treatment of Older Patients With Acute Myelogenous Leukemia
Brief Title: Blood Stem Cell Transplantation for the Treatment of Older Patients With Acute Myelogenous Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2006.065; HUM00006772 (Other: University of Michigan Medical School)
Record Dates: First submitted 2008-02-14; First posted 2008-02-26 (Estimated); Results first posted 2014-07-17 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-03

CONDITIONS: Acute Myelogenous Leukemia
Keywords: AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — fludarabine; Busulfan; Whole-Body Irradiation; Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fludarabine plus Busulfan (CR) (Experimental): Patients in CR will receive a reduced intensity transplant regimen consisting of Fludarabine plus Busulfan (FluBu2).
  Interventions: Drug: Fludarabine; Drug: Busulfan; Radiation: Total Body Irradiation; Procedure: Stem Cell Transplant
- Fludarabine plus Busulfan (PR) (Experimental): Patients in PR will receive a full intensity transplant regimen consisting of Fludarabine plus Busulfan (FluBu4).
  Interventions: Drug: Fludarabine; Drug: Busulfan; Procedure: Stem Cell Transplant

INTERVENTIONS:
Drug: Fludarabine — Fludarabine (40 mg/m2/day x 4 days)
Drug: Busulfan — Busulfan (3.2 mg/m2/day x 2 days or x 4 days).
Radiation: Total Body Irradiation — Patients who receive Busulfan 3.2 mg/m2/day x 2 days and a mismatched allograft (7/8 HLA match) will also receive 200 cGy of total body irradiation (TBI) pre-transplant.
  Arms: Fludarabine plus Busulfan (CR)
Procedure: Stem Cell Transplant — Allogeneic stem cell transplant from related or unrelated donor

SUMMARY:
The prognosis for older individuals with acute myelogenous leukemia (AML) has been historically poor, with 2 year disease-free survival rates < 20% reported. Younger patients with AML in first complete remission are routinely treated using a full intensity (myelo-ablative) chemotherapy followed by a blood stem cell transplant. For the older patient with AML, full intensity therapy transplants have been greatly limited by increased rates of toxic effects related to this type of conditioning regimen. Reduced intensity (non-myeloablative) conditioning regimens have been used in a number of clinical settings, including AML therapy, to lessen the regimen related toxicity in the older patient. Recent data from the University of Michigan Blood and Marrow Transplant Program suggests improved survival for individuals > 55 years in age undergoing reduced intensity, transplants from unrelated donors. This study will investigate the safety and efficacy of this treatment option for older patients with AML, with the primary goal being to improve the survival and lifespan for older patients with AML.

ELIGIBILITY:
Inclusion Criteria:

For Study Registration:

* Age 55 - 70 years.
* Subjects diagnosed with AML (> 20% myeloblasts).

For Proceeding to Transplant:

* Subjects must be in either complete remission (CR) or partial remission (PR) within 14 days prior to admission.
* Subjects must be > 21 days since completion of prior systemic chemotherapy or radiation therapy (including craniospinal XRT), prior to admission .
* Organ function requirements for a reduced intensity (FluBu2) regimen (must be met within 21 days of admission):

  * Cardiac: LV Ejection Fraction > 40% on MUGA or Echocardiogram.
  * Pulmonary: FEV1 and FVC > 40% predicted, DLCO > 40% of predicted.
  * Renal: Serum creatinine < 2.0 mg/dl. Not on hemodialysis or continuous veno-venous filtration (CVVH).
  * Hepatic: serum total bilirubin < 3.0 mg/dl and AST / ALT < 4x ULN
  * Karnofsky > 60%.
* Organ function requirements for a full intensity (FluBu4) regimen (must be met within 21 days of admission):

  * Cardiac: LV Ejection Fraction > 40% on MUGA or Echocardiogram.
  * Pulmonary: FEV1 and FVC > 50% predicted, DLCO (corrected for hemoglobin) > 50% of predicted.
  * Renal: serum creatinine < 2.0 mg/dl. Not on hemodialysis or continuous veno-venous filtration (CVVH)
  * Hepatic: serum total bilirubin < 3.0 mg/dl and AST / ALT < 4x ULN.
  * Karnofsky > 60%.

Exclusion Criteria:

For Study Registration:

* Subjects with M3 AML (FAB classification)

For Proceeding to Transplant:

* Subjects who exhibit signs of progressive disease (> 20% blasts) within 14 days prior to admission for transplant
* Patients with an uncontrolled viral or fungal infection within the prior 28 days.
* Patients who are HIV1 or HIV2 positive.
* Uncontrollable medical or psychiatric disorder

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2007-03; Primary Completion 2013-06 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Yanik, MD, Principal Investigator — University of Michigan Comprehesive Cancer Ctr
Locations (1):
- University of Michigan Cancer Center, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Fludarabine Plus Busulfan: Patients will receive a reduced intensity transplant regimen consisting of Fludarabine (40 mg/m2/day x 4 days) plus Busulfan (3.2 mg/m2/day x 2 days or 3.2 mg/m2/day x 4 days)
  Patients who receive Busulfan at 3.2mg/m2/day x 2 days, and a mismatched allograft (7/8 HLA match), will additionally receive 200 cGy of total body irradiation (TBI) pre-transplant.
  Patients will undergo an allogeneic stem cell transplant from related or unrelated donor.
Period: Overall Study
Arm/Group | Fludarabine Plus Busulfan
Started | 56
Completed | 54
Not Completed | 2
Not completed — Death | 1
Not completed — Patient Declined Transplant | 1

BASELINE CHARACTERISTICS:
Arm/Group | Fludarabine Plus Busulfan
Number analyzed (Participants) | 56
Age, Continuous [Median (Full Range); unit: years] | 61 [55 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 29

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Relapse Free Survival at 1 Year
Description: The primary objective was to determine the 1 year relapse free survival rate (RFS) for individuals > 55 years in age with Acute myeloid leukemia (AML) in Complete Remission (CR) or Partial Remission (PR) who undergo a 7-8/8 HLA- matched unrelated donor transplant using a reduced intensity regimen.
Time Frame: 1 year
Population: 56 patients were enrolled. 54 patients were treated (one died prior to transplant, one did not undergo a transplant) and 4 patients were inevaluable (3 patients were less than 1 year post transplant at the time the abstract was written and 1 failed to engraft).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fludarabine Plus Busulfan
Number analyzed (Participants) | 50
percentage of participants | 56 [43 to 69]

2. Secondary Outcome: Percentage of Participants Alive at 1 Year
Description: One of the secondary objectives was to determine overall survival for patients > 55 years in age with AML undergoing full or reduced transplant with the best available donor.
Time Frame: 1 year
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fludarabine Plus Busulfan
Number analyzed (Participants) | 50
percentage of participants | 58 [46 to 74]

ADVERSE EVENTS:
Arm/Group | Fludarabine Plus Busulfan
Serious Adverse Events (participants affected / at risk) | 21/56
Other Adverse Events (participants affected / at risk) | 16/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fludarabine Plus Busulfan (N=56)
Cardiac ischemia/infarction (Cardiac disorders) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1)
Fever (General disorders) | 3 (4)
Death not associated with CTCAE term (General disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (2)
Hematoma (Vascular disorders) | 1 (1)
Febrile neutropenia (Infections and infestations) | 1 (1)
Blood Infection (Infections and infestations) | 1 (2)
Soft Tissue Infection (Infections and infestations) | 1 (1)
Infection - Other (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 1 (1)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 1 (1)
Confusion (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Mental status (Psychiatric disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Syncope (fainting) (Nervous system disorders) | 2 (2)
Abdomen Pain (Gastrointestinal disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chest/Thorax Pain (Cardiac disorders) | 1 (1)
Syndromes - Other (General disorders) | 1 (1)
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 2 (2)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fludarabine Plus Busulfan (N=56)
Anorexia (Gastrointestinal disorders) | 5 (6)
Mucositis/stomatitis (Gastrointestinal disorders) | 5 (5)
Infection (Infections and infestations) | 4 (7)
Blood Infection (Infections and infestations) | 4 (6)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Thrombosis (vascular access related) (Vascular disorders) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes